CLINICAL TRIAL: NCT00181311
Title: Prospective Investigation of the Incidence of Complications After Vaginal and Abdominal Hysterectomy
Brief Title: Investigation of the Incidence of Complications After Vaginal and Abdominal Hysterectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maasland Hospital (Other)
Other Study IDs: 05-P-26
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2005-08

CONDITIONS: Hysterectomy
Keywords: vaginal hysterectomy; abdominal hysterectomy; complications; physical well being; mental well being
MeSH Terms: conditions — Psychological Well-Being | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: hysterectomy

SUMMARY:
The purpose of this study is to evaluate the short and long term complications after an abdominal or vaginal hysterectomy and to detect the prevalence of occult/subclinical haematomas and vaginal cuff abscesses and the postoperative course of these.

The investigators will also evaluate the physical and mental well being after a hysterectomy with a questionnaire and correlate these results with the occurrence of complications.

DETAILED DESCRIPTION:
Hysterectomy is the most common major gynaecological operation performed worldwide.

The overall average rate of hysterectomy in the United States is 5.6 per 1000 women. There are three different procedures to perform a hysterectomy. The surgery can be approached abdominally, vaginally or as a laparoscopically assisted hysterectomy.

This study will contribute to the improvement of knowledge in short and long term complications and especially the prevalence of occult and subclinical haematomas and vaginal abscesses after abdominal or vaginal hysterectomy. The occurrence of short and long term complications will have an influence on the general well being of the patient. We will also evaluate the physical and mental well being of the patient after a hysterectomy.

After statistical analysis of the study outcome parameters, some conclusions can be drawn for the treatment policy after an abdominal or vaginal hysterectomy to reduce the complication rate and improve the general well being of our patients.

ELIGIBILITY:
Inclusion Criteria:

* Benign indication for undergoing of a hysterectomy
* Written informed consent of the patient

Exclusion Criteria:

* Inability to undergo an operation due to high surgical or anaesthetic risk
* Malignancy as indication for the hysterectomy
* Patients with an enterocele or rectocele and who need prolapse surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2005-08; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Erik Jan Sollie, MD, Study Chair — Maasland Hospital
Locations (1):
- Maasland Hospital, Sittard, Limburg, Netherlands